CLINICAL TRIAL: NCT03188146
Title: Performance of Biochemical Response Criteria and Risk Scoring Systems in Chinese Patients With Primary Biliary Cholangitis (PBC) on Ursodeoxycholic Acid
Brief Title: Performance of Scoring Systems in Chinese Patients With Primary Biliary Cholangitis (PBC) on Ursodeoxycholic Acid
Status: Completed | Type: Observational
Sponsor: Humanity and Health Research Centre (Other)
Collaborators: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: H&H_PBC_01
Record Dates: First submitted 2017-06-08; First posted 2017-06-15 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Primary Biliary Cholangitis (PBC)
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PBC patients with liver biopsy: Ursodeoxycholic acid will be given compliance to the treatment guideline.
  Interventions: Drug: Ursodeoxycholic Acid

INTERVENTIONS:
Drug: Ursodeoxycholic Acid — Standard care of PBC patients

SUMMARY:
Several risk assessment scoring systems have been proposed to assess the therapeutic response and predict long term prognosis in ursodeoxycholic acid (UDCA)-treated primary biliary cholangitis (PBC) patients, in order to risk stratify PBC patients and guide their management. However there scoring systems have not been fully validated in Chinese population. This study is going to compare the prognostic ability of these criteria, validate the overseas scoring systems, develop and validate a new scoring system in a cohort of Chinese PBC patients.

ELIGIBILITY:
Inclusion Criteria:

* With liver biopsy proved PBC

Exclusion Criteria:

* A positive serological test for hepatitis B or C virus,
* Comorbidity of primary sclerosing cholangitis,
* Alcoholic liver disease,
* Hemochromatosis,
* Wilson's disease,
* a1-antitrypsin deficiency
* Presence of complications of cirrhosis (Total bilirubin >100 lmol/L, ascites, variceal haemorrhage and hepatic encephalopathy) on admission.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PBC who are referred to centre of non-infectious liver diseases, Beijing 302 Hospital, Beijing from 2010 will be evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Liver related Death | During follow-up after a year of starting UDCA, an average of 1 year
  Whether the patients die from liver-related causes during the follow-up

SECONDARY OUTCOMES:
Complications of cirrhosis | During follow-up after a year of starting UDCA, an average of 1 year
  Whether the complication of cirrhosis i.e. ascites, hepatic encephalopathy, variceal bleeding occur during the follow-up
Liver transplant | During follow-up after a year of starting UDCA, an average of 1 year
  Whether the patients have liver transplant during the follow-up

CONTACTS AND LOCATIONS:
Overall Officials: George Lau, MD, PhD, Principal Investigator — Humanity and Health Medical Centre
Locations (1):
- Centre of non-infectious liver diseases, Beijing 302 Hospital, Beijing, China., Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided